CLINICAL TRIAL: NCT01229605
Title: Cyclophosphamide and Docetaxel Every 3 Weeks as Neoadjuvant Therapy in Locally Advanced Breast Cancer, A Collaborative Trial
Brief Title: Cyclophosphamide and Docetaxel Every 3 Weeks as Neoadjuvant Therapy in Locally Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not a good fit for the patient population seen at this hospital.
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tufts BR01
Record Dates: First submitted 2010-10-18; First posted 2010-10-28 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Cyclophosphamide and docetaxel every 3 weeks as neoadjuvant chemotherapy
  Interventions: Drug: Cyclophosphamide and docetaxel

INTERVENTIONS:
Drug: Cyclophosphamide and docetaxel — Cyclophosphamide and docetaxel every 3 weeks as neoadjuvant chemotherapy
  Other Names: Cyclophosphamide: Cytoxan; Docetaxel: Taxotere

SUMMARY:
The standard therapy for patients who have locally advanced breast cancer is to receive chemotherapy before surgical removal of tumor. This is called neoadjuvant chemotherapy (NAC). Chemotherapy is used to shrink the tumor before surgery, which sometimes may allow for a smaller portion of the breast to be removed. Receiving chemotherapy before surgery may sometimes also allow for smaller portions of the breast to be removed. Getting chemotherapy prior to surgery may also control any hidden metastatic disease and thereby decrease the risk of cancer relapse. Pre-surgery chemotherapy is a standard management approach for locally advanced breast cancer.

Different combinations of drugs can be used as part of the pre-surgery chemotherapy. The purpose of this study is to determine if using a chemotherapy regimen of TC is effective way to manage locally advanced breast cancer (Stage IIA- IIIB) when the TC is given before surgery. The investigators also hope this study will help us to better understand how the tumor tissue is affected by this combination of chemotherapy drugs.

The TC drug combination is FDA approved for use in treating breast cancer, and it has been shown to be equally effective as other commonly used chemotherapy regimens when used after surgery; but, the TC drug combination has not yet been studied in conjunction with NAC for use before surgery. The investigators will be studying the combination of TC used before surgery as a means of possibly shrinking the tumor.

DETAILED DESCRIPTION:
This is a single-arm, open-label phase II study of cyclophosphamide and docetaxel/taxotere (TC) every 3 weeks in Her2 (-) subjects with locally advanced breast cancer. It is designed to assess (1) the clinical and pathologic response rates to this regimen, as well as its tolerability in this subject population, and (2) the expression of Tiam1 in tumor-associated fibroblasts pre and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older
* Histologically documented adenocarcinoma of the breast, with T2 (T>2.0 cm) N0 or more advanced disease.
* No evidence of metastatic disease.
* Disease must be clinically or radio-graphically measurable or evaluable.
* Incisional or core needle biopsy, yielding sufficient tissue for histologic confirmation of adenocarcinoma, hormone receptor analysis and Her2 testing; and Tiam-1 expression.
* Subjects may have received no prior chemotherapy for breast cancer. Subjects may have received up to 3 months of neoadjuvant hormonal therapy, provided they have been re-staged and are still eligible for this study, and have been off hormonal therapy at least 48 hours.
* Subject must be Her-2 negative.
* Performance status 0-1 by the ECOG scale.
* Baseline laboratory values must be as follows: Absolute granulocyte count: greater than 1400/cells/ml; Platelets: greater than 100,000 cells/ml; Total bilirubin: less than 1.5 mg/dl; Serum ALT: less than 2.5 x institutional upper normal limit; Creatinine: less than 1.6mg/dl; Hemoglobin: greater than 9.0g/dl
* Subjects must be nonpregnant and nonlactating. Subjects of childbearing potential must utilize an effective method of contraception during the study.

Exclusion Criteria:

* Subjects who have received chemotherapy or more than 3 months of neoadjuvant hormone therapy for this cancer.
* Subjects with metastatic disease (disease beyond the breast, axillary nodes and ipsilateral supraclavicular nodes) or inflammatory breast cancer (T4d).
* Subjects with other active cancers, except non-melanoma skin cancers
* Subjects with an active serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment.
* Dementia or significantly altered mental status that would prohibit comprehension of or giving of informed consent.
* Pregnant or breast-feeding women; sexually active, pre-menopausal women not willing to use adequate methods of birth control.
* Subjects who are Her 2 neu positive are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate | 3-4 weeks post-surgery
  The primary outcome measure for this study is the complete response rate for evaluable participants on neoadjuvant chemotherapy with cyclophosphamide and docetaxel. A clinical complete response (cCR) is defined as resolution of all palpable masses.

SECONDARY OUTCOMES:
Change in mean Tiam1 expression levels before and after therapy | Up to 22 weeks
  Descriptive statistic plots and confidence intervals will summarize the observed changes in Tiam1 expression levels before and after therapy. Although primarily descriptive, changes in mean levels pre and post therapy will be tested using the paired t-test or Wilcoxon Signed Ranks Test. Other secondary exploratory analyses will investigate associations between the observed changes in Tiam1 expression and the observed clinical response rate. Regression models will be used to investigate these associations.

CONTACTS AND LOCATIONS:
Overall Officials: John S Nystrom, MD, Principal Investigator — Tufts Medical Center